CLINICAL TRIAL: NCT04622917
Title: Is the Effect of Systemic Steroids Treating Pollen Induced Allergic Rhinitis Mainly Due to a Placebo Effect
Brief Title: Methylprednisolone Injections Treating Birch Pollen Induced Allergic Rhinitis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars Olaf Cardell, Professor, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 791-792
Record Dates: First submitted 2020-10-22; First posted 2020-11-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Rhinitis, Allergic, Seasonal; Hay Fever; Pollen Allergy; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Methylprednisolone; Methylprednisolone Acetate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylprednisolone (Active Comparator): Depo-Medrol (Methylprednisolone) 40 milligrams/milliliter, 2 milliliters as a single dosage
  Interventions: Drug: MethylPREDNISolone 40 Mg/mL Injectable Suspension
- Sodium Chloride (NaCl) (Placebo Comparator): NaCl 0,9 milligrams/milliliter, 2 milliliters as a single dosage
  Interventions: Drug: NaCl 9 MG/ML Injectable Solution

INTERVENTIONS:
Drug: MethylPREDNISolone 40 Mg/mL Injectable Suspension — intramuscular injection
  Other Names: Depo-Medrol
  Arms: Methylprednisolone
Drug: NaCl 9 MG/ML Injectable Solution — Intramuscular injection
  Other Names: Sodium Chloride
  Arms: Sodium Chloride (NaCl)

SUMMARY:
This study evaluates the effect of intramuscular injected methylprednisolone treating birch pollen induced rhinitis compared to placebo.

DETAILED DESCRIPTION:
The study was an interventional single center double-blinded human randomized trial with two groups treated parallel.The first group received an intramuscular injection of Methylprednisolone 40 mg/ml 2ml x 1 as a single dose. The second group received an intramuscular injection of NaCl 0,9 mg/ml 2ml x 1 as a single dose. Symptom score and the use of medication was registered daily during the pollen peak of the season, using an electronic diary. The study was conducted during the spring of 2019.

ELIGIBILITY:
Inclusion Criteria:

* Severe birch pollen induced allergic rhinitis.
* Signed informed consent according to International Council of Harmonisation/Good Clinical Practice, and national/local regulations.
* Women of considered childbearing potential (WOCBP) will only be included after a negative highly sensitive pregnancy test according to CTFG recommendations.

Exclusion Criteria:

* Pregnancy or nursing.
* Autoimmune or collagen disease.
* Cardiovascular disease.
* Hepatic disease.
* Renal disease.
* Cancer.
* Upper airway disease (non-allergic sinusitis, nasal polyposis, chronic obstructive- and restrictive lung disease).
* Medication with a possible side-effect of interfering with the immune response.
* Previous immuno- or chemotherapy.
* Chronic disease.
* Major metabolic disease.
* Alcohol or drug abuse.
* Mental incapability of coping with the study.
* Known or suspected allergy to the study product.
* Suspicion of or confirmed bacterial infection.
* Known allergy to the study drugs, "rescue medication".

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Mean Combined Medical- and Symptom score (CSMS) | 3 weeks
  Daily scoring of rhinoconjunctivitis symptoms (4 questions, 4-point scale. 0= no symptoms and 3=severe symptoms) and use of rescue medication (3-point scale. 0=no medication, 1= oral and/or topical (eyes) non sedative H1 antihistamines (H1A), 2= intranasal corticosteroids with/without H1A) during the birch pollen season.
  CSMS 6-point scale (0=no symptoms and no use of medication, 5= severe symptoms and use of intranasal corticosteroids with/without H1A)
Mean symptom score | 3 weeks
  Daily scoring of rhinoconjunctivitis symptoms (4 questions, 4-point scale. 0= no symptoms and 3=severe symptoms)

SECONDARY OUTCOMES:
Effects on Quality of Life (QoL), SNOT | 3 weeks
  Changes in Sino Nasal Outcome Test 22 (SNOT-22) at trial start, after 1 and 3 weeks respectively.
  22 questions, 6-point scale (0=no change in quality of life and 5=severe reduction in quality of life)
Effects on Quality of Life (QoL), RQLQ | 3 weeks
  Changes in Juniper Rhinitis Quality of Life Questionnaire (RQLQ) at trial start, after 1 and 3 weeks respectively.
  28 questions, 7-point scale ((0=no change in quality of life and 6=severe reduction in quality of life)
Effects on Quality of Life (QoL), ACQ | 3 weeks
  Changes in Asthma Control Questionnaire (ACQ) at trial start, after 1 and 3 weeks respectively.
  5 questions, 7-point scale ((0=no change in quality of life and 6=severe reduction in quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Olaf Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Department of Lung-and Allergy Research, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD of symptoms and use of medication during the trial will be part of the publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Publication planed during 2021.
Access Criteria: The data was published in Scientific reports (found in supplements) 2023
URL: http://www.nature.com/articles/s41598-023-46869-4